CLINICAL TRIAL: NCT03562299
Title: A Prospective, Non-comparative Pilot Clinical Study of a Novel Xenograft Device for Reconstruction of the Anterior Cruciate Ligament.
Brief Title: OrthoPure™ XT Pilot Clinical Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unspecified business decision/strategic reason.
Sponsor: TRX Orthopedics (Industry)
Responsible Party: Sponsor
Organization: Tissue Regenix Ltd (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TRG-A02/0021
Record Dates: First submitted 2018-05-18; First posted 2018-06-19 (Actual); Last update posted 2018-11-21 (Actual); Status verified 2018-11

CONDITIONS: Knee Injuries; Anterior Cruciate Ligament (ACL) Reconstruction
MeSH Terms: conditions — Knee Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Experimental (Experimental): Reconstruction of the Anterior Cruciate Ligament (ACL) using OrthoPure™ XT in patients with a partial or complete tear of the Anterior Cruciate Ligament (ACL)
  Interventions: Device: OrthoPure™ XT

INTERVENTIONS:
Device: OrthoPure™ XT — A decellularized, sterile, single use, xenograft device for reconstruction of the anterior cruciate ligament

SUMMARY:
To evaluate the clinical safety and obtain preliminary effectiveness data for OrthoPure™ XT device in a small group of US patients at 12 and 24 months. The clinical experience obtained from this study will be used to develop a pivotal study for follow up in a larger patient population.

DETAILED DESCRIPTION:
The OrthoPure™ XT device is a decellularized, sterile, single use biological scaffold for use in the treatment of patients with a partial or complete tear of the Anterior Cruciate Ligament (ACL) who require surgical reconstruction of the ACL.

This is a Pilot Safety Study. The primary objective of this study is to evaluate the clinical safety of the OrthoPure™ XT device in a small group of patients that require reconstruction of the Anterior Cruciate Ligament (ACL) due to partial or complete tear of the ACL.

Clinical safety will be analyzed through measurement of immune response (alpha-Gal IgG), blood and urine analysis, incidence of secondary surgical interventions with the treated knee, and the incidence of individual adverse events.

The second objectives of this study are to assess the efficacy endpoints, specifically: improvement in knee stability, function and pain; improvement in patient quality of life and radiographic analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are skeletally mature, as evidenced by closed tibial and femoral epiphyses on x-rays at baseline.
2. Patients who have been diagnosed with a partial or complete tear of the ACL as determined by MRI, require surgical reconstruction of the ACL, and are candidates for ACL surgery.
3. Patients who have passive flexion ≥ 120°, and passive extension on the target knee is the same as the contralateral knee, in the judgment of the Investigator.
4. Patients who have Medial Collateral Ligament (MCL) injury of Grade 2 or less.
5. Patients with osteoarthritis of Grade 2 or less as defined radiographically on the Kellgren-Lawrence (K-L) scale.
6. Patients who are able to give voluntary, written informed consent to participate and have signed an Informed Consent Form specific to this study.
7. Patients who are willing and able to comply with all study procedures including all pre-operative, post-operative and rehabilitation requirements.
8. If female and of child-bearing potential, patients who have a negative urine pregnancy test at Visit 2 and have no intention to become pregnant in the next 24 months.

Exclusion Criteria:

1. Patients with Body Mass Index (BMI) greater than 35 kg/m2.
2. Patients presenting with osteoarthritis of the target knee e.g. International Cartilage Repair Society (ICRS) Grade III or higher as determined by their baseline MRI scan.
3. Patients who have had previous ACL reconstruction on the target knee.
4. Patients who have had any other type of surgical procedure on the target knee in the 3 months prior to Visit 1.
5. Patients with ligament instability, osteoarthritis greater than Grade 2 or a current ACL injury in the contralateral knee.
6. Patients with a complete or partial Lateral Collateral Ligament (LCL) tear or Posterior Cruciate Ligament (PCL) tear on the target knee.
7. Patients with meniscal repairs and tears requiring more than one third (1/3) removal of the meniscus on the target knee as determined during knee arthroscopy.
8. Patients who have an active systemic infection, or an active local infection in or near the target knee, or have a previous history of joint infection.
9. Patients who are participating concurrently in another clinical trial, or have participated in a clinical trial within the last 90 days, or intend to during the course of the study.
10. Patients who have previously been implanted with any type of xenograft device.
11. Patients with known immunodeficiency including patients who are receiving or have received corticosteroids, immunosuppressants, immunostimulating agents or radiation therapy within 6 months of Visit 1.
12. Patients who have conditions that may be exacerbated by, or may interfere with the results of the skin prick test.
13. Patients with significant comorbidities or conditions associated with high risk for surgical or anesthetic survival (e.g. renal failure, peripheral vascular disease, unstable cardiac disease, poorly controlled diabetes, immunosuppression, etc.).
14. Patients with active neoplastic disease.
15. Patients with known allergy to mammalian meat, porcine products or a religious objection to the use of implanted porcine material.
16. Patients with current drug or alcohol abuse, or a history of the same within the last 6 months.
17. Patients with local circulatory problems, (e.g. thrombophlebitis and lymphedema).
18. Patients with any mental or psychological disorder that would impair their ability to complete the study questionnaires.
19. Patients with any medical condition or other circumstances that might interfere with their ability to return for follow-up visits in the judgment of the Investigator, including any systemic illness, neuromuscular, neurosensory, or musculoskeletal deficiency that would render the patient unable to perform appropriate postoperative rehabilitation.
20. Any condition which, in the judgment of the Investigator, would preclude adequate evaluation of device's safety and performance.

    -

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2018-07 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Assessment of anti-Gal IgG antibody levels | profile up to 24 months
  Blood sample collection for measurement of immune response
Measurement of serum chemistry | up to 24 months
  Blood sample analysis
Incidence of secondary surgical interventions (SSIs) | up to 24 months
  The frequency and seriousness of any secondary surgical interventions will be assessed.
Incidence of individual Adverse Events | up to 24 months
  The frequency and seriousness of any adverse events or adverse device.effects will be assessed.

SECONDARY OUTCOMES:
Improvement in knee stability - Pivot Shift Test | 3, 6, 12 and 24 months
  Measured by the assessment of change in the anterior cruciate instability in the treated knee
Improvement in knee stability - Lachman test | 3, 6, 12 and 24 months
  Measured by clinical examination of the treated knee (assessment of anterior translation), more than about 2 mm of anterior translation compared to the normal opposite knee suggests an ACL tear
Improvement in knee stability - Anterior Drawer Test | 3, 6, 12 and 24 months
  Clinical assessment of the treated knee, an increased amount of anterior tibial translation compared with the opposite, normal knee can indicate an ACL tear. If the tibia pulls forward or backward more than normal, the test is considered positive
Arthrometric measurement of knee joint laxity | 3, 6, 12 and 24 months
  Comparison of the side-to-side differences in mm between the treated knee and the opposite normal knee using an arthrometric ligament testing device
Improvement in pain and function of the knee measured by questionnaires | 6,12 and 24 months
  Patient's subjective score of 1 to 100 points, with 100 implying the best results and 1 the worse results
Evidence of integration of the investigational product | 3, 6, 12 and 24 months
  MRI assessments
Improvement in quality of life | 3, 6, 12 and 24 months
  A questionnaire on the self-assessment of health condition reflecting the physical condition and mental health
Assessment of investigational device usability | Day 0
  Surgeon assessment of the device (questionnaire), rate from excellent to poor
Assessment on Bone Tunnel Position | 2 weeks, 6 Months
  To be assessed via X Ray

CONTACTS AND LOCATIONS:
Overall Officials: Tom Carter, Principal Investigator — St. Joseph's Outpatient Surgery Center; Jack Farr, Principal Investigator — OrthoIndy Hospital South; David Caborn, Principal Investigator — Jewish Hospital and St. Mary's Healthcare
Locations (3):
- United States (3):
  - St.Joseph's Outpatient Surgery Center, Phoenix, Arizona
  - OrthoIndy Hospital South, Greenwood, Indiana
  - Jewish Hospital, Louisville, Kentucky